CLINICAL TRIAL: NCT00458718
Title: Single Country, Double-Blind, Randomized, 2-Arm, Parallel-Group Study, Evaluating Efficacy and Safety of Rimonabant 20 mg OD, With/Without Association of Nicotine Patch, as Aid to Smoking Cessation During 9-Week Period
Brief Title: Efficacy and Safety of Rimonabant as an Aid to Smoking Cessation With or Without Nicotine Patch
Acronym: CIRRUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC4798
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Smoking Cessation
Keywords: abstinence; nicotine patch
MeSH Terms: conditions — Smoking Cessation | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: rimonabant (SR141716)

SUMMARY:
The primary objective is to compare the efficacy of rimonabant 20 mg OD fixed dose plus nicotine patch 21 mg OD with the combination rimonabant 20 mg OD fixed dose plus placebo patch on abstinence from smoking in cigarette smokers motivated to quit.

Secondary objectives are to evaluate the clinical and biological safety of rimonabant associated with nicotine replacement therapy during a 9-week treatment period and to evaluate the effect of the combination on weight and craving.

ELIGIBILITY:
Inclusion Criteria:

* Smokers smoking at least 15 cigarettes/day as a mean within the 2 months preceding the screening visit
* Motivated to quit with a score greater than or equal to 6 on the ten-point Motivation Scale

Exclusion Criteria:

* non tobacco cigarettes consumption
* chronic use of marijuana
* pregnancy
* breastfeeding
* any clinically significant disease that might interfere with the efficacy or safety evaluation of the study drug
* Concomitant use of drugs as an aid to smoking cessation or that might induce weight change

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2004-09; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Prolonged abstinence from smoking during the last 4 weeks of treatment reported by the subject and confirmed by exhaled carbon monoxide (CO) measurements

SECONDARY OUTCOMES:
Efficacy: mean change of the total score of Questionnaire on Smoking Urges (QSU) brief scale, categorical change in body weight in subjects with Body Mass Index lower than 30 kg/m² at baseline who achieve prolonged abstinence
Safety data

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States

REFERENCES:
- [Derived] Rigotti NA, Gonzales D, Dale LC, Lawrence D, Chang Y; CIRRUS Study Group. A randomized controlled trial of adding the nicotine patch to rimonabant for smoking cessation: efficacy, safety and weight gain. Addiction. 2009 Feb;104(2):266-76. doi: 10.1111/j.1360-0443.2008.02454.x. PMID 19149823